CLINICAL TRIAL: NCT04529733
Title: Evaluation of the IB10 Sphingotest PCT+ in a Point-of-Care Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nexus DX (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B10-08
Record Dates: First submitted 2020-08-14; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: IB10 sphingotest PCT+ — Whole blood in EDTA for procalcitonin POC testing on IB10 sphingotest PCT+ device

SUMMARY:
To establish the equivalence of IB10 sphingotest PCT+ measurements in point-of-care settings such as emergency rooms or intensive care units, with corresponding procalcitonin measurements obtained in a reference or clinical laboratory using a comparative assay, with respect to the same subset of human EDTA plasma specimens.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to provide written informed consent
* Subject is 18 years of age or older
* Subject is presenting with symptoms suggestive of bacterial infection
* Subject is presenting with two or more of the following symptoms suggestive of systemic inflammatory response syndrome (SIRS):

  * Body temperature less than 36°C (96.8°F) or greater than 38°C (100.4°F);
  * Heart rate greater than 90 beats per minute;
  * Respiratory rate greater than 20 breaths per minute, or an arterial partial pressure of carbon dioxide (pCO2) less than 4.3 kPa (32 mmHg);
  * White blood cell count less than 4,000 cells/mm3 (4 x 109 cells/L) or greater than 12,000 cells/mm3 (12 x 109 cells/L);
  * A normal white blood cell count with the presence of greater
  * than 10% immature neutrophils.

Exclusion Criteria:

* Subjects less than 18 years of age;
* Subjects who do not present with a minimum of two symptoms suggestive of SIRS, as defined above
* Subjects unable or unwilling to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
To establish the equivalence of IB10 sphingotest PCT+ measurements in point-of-care settings, with corresponding procalcitonin measurements obtained in a ref or clinical laboratory using a comparative assay, with respect to the same EDTA plasma specimens | 1 day
  Method comparison
To establish the equivalence of IB10 sphingotest PCT+ measurements in EDTA whole blood and plasma specimens, as obtained in point-of-care settings as defined above | 1 day
  Method comparison
To establish equivalence of IB10 sphingotest PCT+ measurements in fresh EDTA plasma specimens and frozen EDTA plasma specimens | 24 hours
  in vitro stability
To establish the precision of IB10 sphingotest PCT+ measurements in point-of-care setting with respect to frozen EDTA plasma specimens | 1 day
  Point of Care precision Testing
To establish the in vitro stability of EDTA whole blood and plasma speciments with respect to procalitonin concentrations as measured by the of IB10 sphingotest PCT+ test. | 1 day
  in vitro stability

IPD SHARING:
Plan to Share IPD: No